CLINICAL TRIAL: NCT00557947
Title: Multi-centre Study to Show Equivalence of Prineo (Dermabond Protape) to Intradermal Sutures for Skin Closure of Full-thickness Surgical Incisions
Brief Title: Prineo (Dermabond Protape) Versus Sutures for Full-thickness Surgical Incisions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06CS005
Record Dates: First submitted 2007-11-09; First posted 2007-11-14 (Estimated); Results first posted 2012-07-19 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-06

CONDITIONS: Surgical Incisions
Keywords: Abdominoplasty; Body Lift; Plastic Surgery; Skin Closure; Wound Healing; Dermabond
MeSH Terms: conditions — Surgical Wound | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Dermabond Protape-Incision segments are randomized & patient is own control
  Interventions: Device: Dermabond Protape (Prineo)
- II (Active Comparator): Intradermal Suture - Incision segments are randomized & patient is own control. Investigator selected suture on the basis of standard local practice.
  Interventions: Device: Suture

INTERVENTIONS:
Device: Suture — intradermal and topical suturing
  Other Names: Investigator selected the intradermal suture per standard local practice.
  Arms: II
Device: Dermabond Protape (Prineo) — cyanoacrylate and pressure sensitive adhesive mesh - topical skin adhesive
  Other Names: Prineo
  Arms: I

SUMMARY:
This is a prospective, controlled, randomized, multi-center clinical study of up to 80 subjects with full thickness surgical incisions. Each incision included in the study will be segmented into two halves; each half will be randomized to receive final skin closure with either Prineo (DERMABOND PROTAPE) or intradermal sutures. Subjects will be evaluated post-operatively at 24 hours (± 6 hours), 7 days (± 1 day), 12 - 25 days, and 90 days (± 10 days).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Be in good general health in the opinion of the Investigator with no conditions that would significantly impact wound healing as determined by medical history and review of recent concomitant medications;
* Be scheduled for at least one full thickness surgical incision of at least 20cm in length as part of elective abdominoplasty or body lift procedures, requiring the placement of sutures in the superficial fascia and subcutaneous tissue to relieve skin tension prior to final skin closure;
* Be willing to follow instructions for incision care as instructed by the investigator, and refrain from swimming or soaking in a tub during the first 12 - 25 days of the study;
* Agree to return for all follow-up evaluations specified in this protocol [7 days (± 1 day), 12 - 25 days, and 90 days (± 10 days)], six (± 1 month) and twelve months (± 1 month)];
* Agree not to schedule any additional elective surgical procedures that involve an incision that is randomized for inclusion in this study, until their participation in this study is complete; and
* Sign the informed consent.

Exclusion Criteria:

* Have peripheral vascular disease;
* Have insulin dependent diabetes mellitus;
* Be known to have a blood clotting disorder;
* Be receiving antibiotic therapy for pre-existing condition or infection;
* Be known to be HIV-positive or otherwise immunocompromised;
* Have known personal or family history of keloid formation or hypertrophy;
* Be currently taking systemic steroids;
* Have known or suspected allergy or sensitivity to cyanoacrylate, formaldehyde, tapes or adhesives
* Have incision type or location known to have an incidence of cyanosis or other healing abnormalities; and
* Be participating in any current clinical trial or have participated in any clinical trial within 30 days of enrolment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Colquhoun, MD, Study Director — Pleiad Devices
Locations (5):
- UZ, Ghent, Belgium
- Germany (2):
  - Dreifaltigkeits-Krankenhaus, Cologne
  - Markus Krankenhaus, Frankfurt
- Akademikliniken, Stockholm, Sweden
- Mid Essex Hospital, Broomfield, Essex, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the general population undergoing elective surgical procedures for body contouring.
Groups:
- Dermabond Protape/Suture: Dermabond Protape-Incision segments are randomized & patient is own control. Incision segments are randomized such that each patient receives Dermabond Protape to close one side of the incision and Intradermal Sutures to close the other side of the incision. Protape is supplied as a single use mesh device with sufficient adhesive to saturate mesh. Sutures were not supplied.
Period: Overall Study
Arm/Group | Dermabond Protape/Suture
Started | 83
Completed | 83
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dermabond Protape/Suture
Number analyzed (Participants) | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 74
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 6
Region of Enrollment [Number; unit: participants]
  Belgium | 22
  Germany | 36
  United Kingdom | 20
  Sweden | 5

OUTCOME MEASURES:

1. Primary Outcome: Continuous Apposition of the Skin Edges Without Wound Dehiscence or Re-closure as Measured by the Upper Limit of 95% Confidence Interval in Proportion of Successes for Each Groups.
Description: Equivalence is demonstrated if the upper limit of the 95% confidence interval (when subtracting the percentage of DERMABOND PROTAPE successful subjects from the percentage of INTRADERMAL SUTURE successful subjects) does not exceed 12%.
Time Frame: 12-25 days post-operation
Population: The primary analysis is based upon intent to treat population.
Measure: Number; unit: Participants
Groups:
- Dermabond Protape: Dermabond Protape-Incision segments are randomized & patient is own control
- Suture: Suture - Incision segments are randomized & patient is own control.
Arm/Group | Dermabond Protape | Suture
Number analyzed (Participants) | 83 | 83
Participants | 74 [0 to 10.9] | 78 [0 to 10.9]
Statistical Analysis 1: Comparison: Dermabond Protape vs Suture; Test type: Non-Inferiority or Equivalence — Equivalence is demonstrated if the upper limit of the 95% confidence interval (when subtracting the percentage of DERMABOND PROTAPE successful subjects from the percentage of INTRADERMAL SUTURE successful subjects) does not exceed 12%; p = 0.2188, McNemar; difference proportions of successes (%) = 4.8, 95% CI 2-sided [-0.0 to 10.9] — The level of significance for statistical testing was 0.05 for this study

2. Secondary Outcome: Time Required to Close the Final Skin Layer
Description: Time to close final skin layer for each incision segment.
Time Frame: Intraoperative
Population: The analysis is based upon the Intent To Treat population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Dermabond Protape | Suture
Number analyzed (Participants) | 83 | 83
minutes | 1.46 (0.96) | 6.65 (4.02)
Statistical Analysis 1: Comparison: Dermabond Protape vs Suture; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Cosmetic Outcome
Description: Modified Hollander Cosmesis Scale overall outcome score in which a score of 0 corresponds to a good outcome versus a 1-6 to a poor outcome. The proportions of incisions with good outcomes were then compared to those with poor outcomes.
  Reference: Hollander JE, Singer AJ, Valentine S, Thode HC Jr, Henry MC. Wound registry:development and validation. Ann Emerg Med. 1995;25:675-85.
Time Frame: 90 days post-procedure
Population: There were 50 participants who consented to and ultimately attended follow-up visits for evaluation of cosmetic outcome.
Measure: Number; unit: Incisions with good outcome
Arm/Group | Dermabond Protape | Suture
Number analyzed (Participants) | 50 | 50
Incisions with good outcome | 33 | 37
Statistical Analysis 1: Comparison: Dermabond Protape vs Suture; Test type: Superiority or Other; p = 0.3877, McNemar

4. Secondary Outcome: Cosmetic Outcome
Description: as for outcome 3
Time Frame: 6 months
Population: There were 50 participants who consented to and ultimately attended all follow-up visits for evaluation of cosmetic outcome.
Measure: Number; unit: Incisions with good outcomes
Arm/Group | Dermabond Protape | Suture
Number analyzed (Participants) | 50 | 50
Incisions with good outcomes | 30 | 32
Statistical Analysis 1: Comparison: Dermabond Protape vs Suture; Test type: Superiority or Other; p = 0.7539, McNemar

5. Secondary Outcome: Cosmetic Outcome
Description: as for outcome 3
Time Frame: 12 month
Population: There were 49 participants who consented to and ultimately attended all follow-up visits for evaluation of cosmetic outcome.
Measure: Number; unit: Incisions with good outcome
Arm/Group | Dermabond Protape | Suture
Number analyzed (Participants) | 49 | 49
Incisions with good outcome | 33 | 32
Statistical Analysis 1: Comparison: Dermabond Protape vs Suture; Test type: Superiority or Other; p = 1.0000, McNemar

ADVERSE EVENTS:
Groups:
- Unrelated: Reported events per local regulatory requirements but not related to either device or procedure.
Arm/Group | Dermabond Protape | Suture | Procedure | Unrelated
Serious Adverse Events (participants affected / at risk) | 3/83 | 3/83 | 11/83 | 3/83
Other Adverse Events (participants affected / at risk) | 16/83 | 16/83 | 24/83 | 7/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dermabond Protape (N=83) | Suture (N=83) | Procedure (N=83) | Unrelated (N=83)
Wound Dehiscence (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Subject experienced wound dehiscence due to an infection. No action taken regarding device. The event was not related to the sutures, possibly related to the DERMABOND PROTAPE, and definitely related to the procedure.
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The subject experienced an infection and seroma. There was no action taken regarding the study device, The infection was classified as not related to either the sutures or the DERMABOND PROTAPE, but was definitely related to the procedure.
Seroma (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The subject experienced an infection and seroma. There was no action taken regarding the study device, The seroma was classified as not related to either the sutures or the DERMABOND PROTAPE but was definitely related to the procedure.
Wound Necrosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Subject experienced wound necrosis requiring surgical treatment. No action required with respect to device. The event was classified as not related to INTRADRERMAL SUTURES or the DERMABOND PROTAPE, but was definitely related to the procedure.
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Subject experienced infection and seroma. No action was taken with device. The infjection was assessed as possibly related to sutures, not related to DERMABOND PROTAPE, and definitely related to the procedure.
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — The subject experienced an infection and seroma. No action was taken regarding the study device for either device. The seroma was classified as possibly related to sutures, not related to DERMABOND PROTAPE, and definitely related to the procedure.
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Subject experienced chest pain. No action was taken with study device. The event was classified as not related to sutures, DERMABOND PROTAPE, or the procedure.
Metastic Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The subject died of metastatic breast cancer. In the opinion of the investigator, the event was classified as not related to either the study device/procedure.
Procedural Complication (requiring removal of skin flap) due to congestion of blood supply (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Subject required required removal of the flap due to congestion of blood supply.There was no action taken regarding study device. Te event was classified as not related to the suture OR DERMABOND ROTAPE, but definitely related to the procedure.
Fluid Overload (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — During surgery, the subject experienced fluid overload (fluid induced respiratory depression). No action was taken with study device. The event was classified as not related to sutures or DERMABOND PROTAPE, and definitely related to the procedure
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The subject experienced hematoma and dehiscence. No action was taken with device with respect to hematoma. The event was no related to sutures or DERMABOND PROTAPE, and definitely related to the procedure.
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The subject experienced hematoma and dehiscence. No action was taken with device with respect to dehiscence. The event was no related to sutures or DERMABOND PROTAPE, and definitely related to the procedure.
Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Subject experienced hematoma, infection and dehiscence following treatment. The infection was classified as possibly related to sutures and DERMABOND PROTAPE and as definitely related to the procedure.
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Subject experienced hematoma, infection and dehiscence following treatment. The infection was classified as related to sutures, possibly related to DERMABOND PROTAPE, and definitely related to the procedure
Hematoma (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Subject experienced hematoma, infection and dehiscence following treatment. No action was taken with devices for the events. The hematoma was classified as possibly related to sutures and DERMABOND PROTAPE, and definitely related to the procedure.
Wound Infection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — The subject experienced wound infection (DERMABOND PROTAPE side). No was action taken regarding the study device. The event was classified as not related to sutures, definitely related to DERMABOND PROTAPE, and possibly related to the procedure.
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The subject experienced arrhythmia (Tachycardia) and breast abscess. No action taken regarding the study device with respect to arrythmia. The event was classified as not related to sutures or DERMABOND PROTAPE, and possibly related to the procedure.
Breast Abcess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The subject experienced arrhythmia (Tachycardia) and breast abscess. No action taken regarding the study device with respect to abscess. The abscess was classified as not related to the sutures or DERMABOND PROTAPE, or the procedure.
Necrosis (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — The subject experienced necrosis (blood supply problem to breast reconstruction) requiring device removal.The event was classified as possibly related to sutures, not related to DERMABOND PROTAPE, and definitely related to procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Dermabond Protape (N=83) | Suture (N=83) | Procedure (N=83) | Unrelated (N=83)
Pain (General Disorders) (General disorders) | 16 (16) | 16 (16) | 19 (19) | 0 (0) — Pain at application site.
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (83) | 0/0 (0) — Nausea experienced following surgery.
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (5) | 0/0 (0) — Insomnia experienced following surgery.
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 6 (6)
Procedure Pain (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 5 (5) | 0/0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of this study include the fact that the patient served as her own control. Additionally, as in many device studies, because of the obvious difference in the investigated and the control devices, blinding was limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less